CLINICAL TRIAL: NCT03097757
Title: Randomized Controlled Trial of Ultrasound Guidance for Reduction of Pediatric Forearm Fractures
Brief Title: Trial of Ultrasound Guidance for Reduction of Pediatric Forearm Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit patients for this study due to time constraints and personnel limitations.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2016-6637
Record Dates: First submitted 2017-03-25; First posted 2017-03-31 (Actual); Results first posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Forearm Fracture; Ultrasound
Keywords: Ultrasound; Forearm Fracture Reduction; Pediatric Emergency Department

STUDY DESIGN:
Intervention Model Description: Prospective randomized, controlled, single blinded study
Who Masked: Outcomes Assessor
Masking Description: The orthopedic surgeon reading the x-rays and determining the degree of angulation and displacement will be blinded to all patient characteristics and to the patient's group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Fracture reduction without ultrasound (Active Comparator): Fracture reduction as per standard of care involves closed fracture reduction without real-time imaging, or with c-arm or portable x-ray. Closed reduction of a fractured bone. Closed reduction is a procedure to set (reduce) a broken bone without surgery. This allows the bone to grow back together. It works best when it is done as soon as possible after the bone breaks.
  Interventions: Procedure: Standard of care fracture reduction
- Fracture reduction with ultrasound (Experimental): Ultrasound guided Fracture reduction involves closed fracture reduction with the use of real-time ultrasound imaging, prior to, during and after the reduction procedure. C-arm or portable x-ray may also be used as an adjunct.
  Interventions: Radiation: Ultrasound - guided fracture reduction; Procedure: Standard of care fracture reduction

INTERVENTIONS:
Radiation: Ultrasound - guided fracture reduction — Ultrasound will be used as a real-time imaging modality to guide forearm fracture reduction.
  Arms: Fracture reduction with ultrasound
Procedure: Standard of care fracture reduction — Closed reduction of a fractured bone.

SUMMARY:
The primary objective of this study is to assess the utility of ultrasound guidance in the closed reduction of pediatric forearm fractures in the pediatric emergency department. The investigators will compare post-reduction radiologic outcomes between the experimental group (ultrasound guided closed forearm fracture reduction) and control group (standard of care blinded closed forearm fracture reduction) to determine if there is a difference in the number of adequate reductions between groups.

Secondary objectives include comparing provider satisfaction with the reduction procedure, number of patients requiring repeat reductions, time for reduction, number of patients requiring operative repair after reduction, with the reduction procedure and comparison between post-reduction ultrasound and x-ray interpretation.

DETAILED DESCRIPTION:
This will be a prospective randomized, controlled, single blinded study that will take place at the Children's Hospital at Montefiore (CHAM) in the Pediatric Emergency Department (PED). Patients who present to the PED, are confirmed to have a forearm fracture requiring closed reduction in the PED and meet the inclusion/exclusion criteria will be eligible for the study. The decision to perform a closed reduction procedure in the PED will be made by the consulting orthopedic surgeon who will perform the procedure. All eligible patients' pain will be reassessed and managed as necessary as per standard of care The eligible patient or parent/guardian will be approached by the treating physician or consulting orthopedic resident for written consent. Written assent will be obtained from minors older than 7 years of age. After enrollment into the study, patients will be randomized to either the experimental group (ultrasound guided fracture reduction) or control group (standard of care forearm fracture reduction without real-time imaging). Allocation of patients to intervention and control arms will be accomplished by a computer-generated permuted block randomization scheme.

Consulting orthopedic residents will be trained to perform musculoskeletal sonography for this study and will be considered study-trained physicians. All patients will undergo procedural sedation and/or pain management for closed reduction as per standard of care in the PED. The medication used for sedation and/or pain will be determined by the treating Pediatric Emergency Medicine (PEM) physician. Study patients that are randomized to the ultrasound guided group will undergo a point-of-care ultrasound, performed by a study trained physician using a Sonosite Edge ultrasound machine with an L38 linear 10-5 Megahertz (MHz) transducer probe.

Prior to the reduction procedure in patients randomized to the experimental group, ultrasound images of the fracture site will be obtained and the maximum degree of displacement will be measured. Both longitudinal and transverse views of the injured area will be obtained. The trained physician will then perform real-time ultrasound imaging as needed during the closed reduction procedure. Once the orthopedic resident obtains optimal alignment, and prior to casting, a post-reduction ultrasound image will be obtained and the angle of displacement will again be measured. All ultrasounds performed prior to and after the reduction will be recorded, and the images obtained will include video clips of the ultrasound as well as a saved still picture of the best image of the suspected fracture site. The study-trained physician who performed the ultrasound will then record his/her findings on the data collection form immediately after the procedure and prior to reviewing plain radiographs.

In general, the majority of reduction procedures performed in the PED are done without the use of any real time imaging, some orthopedic surgery residents employ the use of the c-arm (fluoroscopy) and/or a portable x-ray machine during the reduction procedure. At his/her discretion, the orthopedic resident may use either of these modalities in both the ultrasound and control group as per standard of care in the PED. The use of these modalities will be recorded.

After the reduction procedure in the ultrasound group and prior to reviewing the post reduction x-ray, the orthopedic resident will complete a brief questionnaire. Patients in both groups will then undergo a post-reduction x-ray. Based on the degree of displacement on the x-ray, the orthopedic surgeon will determine whether the patient needs a repeat reduction, as per routine standard of care. If a repeat reduction is required, the treating physician can choose to use ultrasound at his/her discretion. The angle of displacement will be measured on the post-reduction x-ray by an orthopedic surgeon. Additionally, the angle of displacement measured on the post-reduction ultrasound will be measured and compared to the angle of displacement on the post-reduction x-ray. An expert sonographer will review cases where the ultrasound and x-ray results do not correlate.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to the Pediatric Emergency Department (PED) with a confirmed displaced forearm fracture that will require reduction by orthopedic surgery in the PED will be eligible for inclusion in this study.

Exclusion Criteria:

1. Patients with open fractures.
2. Patients with neurovascular compromise.
3. Unstable patients with life-threatening injuries who require ongoing resuscitation.

Max Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joni Rabiner, MD, Principal Investigator — Columbia University
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fracture Reduction Without Ultrasound | Fracture Reduction With Ultrasound
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fracture Reduction Without Ultrasound | Fracture Reduction With Ultrasound | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Comparing Rate of Reduction Between the Experimental and Control Arm/Group
Description: To compare the number of patients requiring repeat reduction procedure between the experimental group (ultrasound guided fracture reduction) and control group (standard of care forearm fracture reduction).
Time Frame: From initiation of bone setting procedure, an average of 10-20 minutes
Population: Data were not collected/aggregated and therefore data analysis was not conducted as only 4 patients were enrolled into the study (2 into each Arm/Group). Per protocol, the plan was to enroll 56 patients into each of the two study Arms/Groups (n=112). Allocation of patients into each arm was to have been conducted by a computer-generated permuted block randomization scheme to mitigate experimental error contributed by inexperience using the ultrasound guidance at the start of the study.
Arm/Group | Fracture Reduction Without Ultrasound | Fracture Reduction With Ultrasound
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Compare Provider Satisfaction With the Reduction Procedure Between the Experimental and Control Arm/Group
Description: Based on a questionnaire asking:
  For the experimental Arm/Group (fracture reduction with ultrasound):
  1. Ease of fracture reduction on 5-point scale (ranging from 1 = easy to 5 = very difficult)
  2. Ease of using ultrasonography on 5-point scale (ranging from 1=easy to 5 = very difficult)
  3. Was ultrasound helpful in completing fracture reduction? Assessed on a trinary option of a) yes, b) no, c) uncertain
  For the Control Arm/Group (fracture reduction without ultrasound):
  1. Ease of fracture reduction on 5-point scale (ranging from 1 = easy to 5 = very difficult)
  2. Do you think real-time imaging would have been helpful for this reduction? Assessed based on a trinary option of a) yes, b) no, c) uncertain
Time Frame: After completing the bone setting procedure and validation via ultrasound, an average of 2 minutes
Population: as for outcome 1
Arm/Group | Fracture Reduction Without Ultrasound | Fracture Reduction With Ultrasound
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Adequacy of Reduction Based on a Composite Assessment of Degree of Angulation and Displacement
Description: To compare the adequacy of reduction between the experimental and control Arm/Group by a composite assessment of the degree of angulation and displacement on post reduction x-rays. The acceptable degree of angulation will be the same in both Arms/Groups. The acceptable degree of angulation based on age is less than 20 degrees' angulation for patients younger than 10 years of age and less than 10 degrees' angulation for patients older than 10 years of age.
  To compare the adequacy of reduction between the experimental and control Arm/Group by measuring and comparing the degree of displacement on the post reduction x-rays.
Time Frame: From initiation of bone setting procedure, an average of 10-20 minutes
Population: as for outcome 1
Arm/Group | Fracture Reduction Without Ultrasound | Fracture Reduction With Ultrasound
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Reduction
Description: To compare the time for the fracture reduction procedure between the experimental and control Arm/Group.
Time Frame: From initiation of bone setting procedure, an average of 10-20 minutes
Population: as for outcome 1
Arm/Group | Fracture Reduction Without Ultrasound | Fracture Reduction With Ultrasound
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Operative Repair
Description: To compare the number of patients requiring operative repair after reduction between the experimental and control Arm/Group.
Time Frame: From initiation of bone setting procedure, an average of 10-20 minutes
Population: as for outcome 1
Arm/Group | Fracture Reduction Without Ultrasound | Fracture Reduction With Ultrasound
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Post-Reduction Ultrasound Comparison
Description: To compare the post-reduction ultrasound, including measurement of degree of angulation and displacement, for each patient.
Time Frame: From initiation of bone setting procedure, an average of 10-20 minutes
Population: as for outcome 1
Arm/Group | Fracture Reduction Without Ultrasound | Fracture Reduction With Ultrasound
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Post-Reduction X-ray Interpretation
Description: To compare the post-reduction x-ray interpretation, including measurement of degree of angulation and displacement on the x-raym for each patient.
Time Frame: From initiation of bone setting procedure, an average of 10-20 minutes
Population: as for outcome 1
Arm/Group | Fracture Reduction Without Ultrasound | Fracture Reduction With Ultrasound
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for the duration of their emergency department visits, i.e., approximately 1-2 hours post procedure.
Arm/Group | Fracture Reduction Without Ultrasound | Fracture Reduction With Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects recruited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT03097757/Prot_SAP_001.pdf